CLINICAL TRIAL: NCT04728698
Title: Treatment of COVID-19-Induced Acute Respiratory Distress: A Phase 2 Study of Intravenous Administration of Allogeneic Adipose-Derived Mesenchymal Stem Cells
Brief Title: Study of Intravenous Administration of Allogeneic Adipose-Derived Mesenchymal Stem Cells for COVID-19-Induced Acute Respiratory Distress
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Replaced by a different protocol.
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSC-COV-201
Record Dates: First submitted 2021-01-26; First posted 2021-01-28 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Covid19; ARDS
Keywords: covid-19; ARDS
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- COVI-MSC (Experimental): Allogeneic culture-expanded adipose-derived mesenchymal stem cells (MSCs)
  Interventions: Drug: COVI-MSC
- Placebo (Placebo Comparator): Excipient
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: COVI-MSC — 1 x 10^6 MSCs/kg or 1.5 x 10^6 MSCs/kg, depending on CRP level
  Arms: COVI-MSC
Drug: Placebo — Equivalent volume of placebo will be administered
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized controlled, multicenter study to assess the safety and efficacy of COVI-MSC in the setting of current standard of care (SOC) treatments for COVID-19 infection in hospitalized subjects with ARD/ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Provides informed consent
* Has laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR) or other commercial or public health assay in any specimen
* 3. Is hospitalized with COVID-19-induced ARD or ARDS (any severity) with a PaO2/FiO2 ≤300. The PaO2/FiO2 may be estimated from pulse oximetry or determined by arterial blood gas
* Requires oxygen supplementation at screening
* Is willing to follow contraception requirements

Exclusion Criteria:

* Current standard of care treatments for COVID-19 appear to be working and the subject is clinically improving
* A previous MSC infusion unrelated to this trial
* Have any of the following medical conditions:

  * Cardio-pulmonary resuscitation within 14 days of randomization
  * Uncontrolled or untreated symptomatic arrhythmias. Exception: Subjects with controlled, asymptomatic atrial fibrillation during screening may enroll
  * Myocardial infarction within the last 6 weeks
  * Congestive heart failure (NYHA Grade 3 or 4)
  * Pulmonary hypertension (WHO Class III/IV)
  * Currently receiving extracorporeal life support or membrane oxygenation (ECLS/ECMO)
  * Alanine aminotransferase (ALT) ≥ 5x upper limit of normal (ULN)
  * Relevant renal impairment (eGFR < 50 mL/min)
  * Any significant medical condition, laboratory abnormality or psychiatric illness that in the investigator's opinion would interfere or prevent the subject from safely participating in the study
* Pregnant or breast feeding or planning for either during the study
* Suspected uncontrolled active bacterial, fungal, viral, or other infection (aside from infection with COVID-19)
* History of a splenectomy, lung transplant or lung lobectomy;
* Concurrent participation in another clinical trial involving therapeutic interventions (observational study participation is acceptable).
* Expected survival or time to withdrawal of life-sustaining treatments expected to be < 7 days.
* Do Not Intubate order;
* Home mechanical ventilation (noninvasive ventilation or via tracheotomy) except for continuous positive airway pressure or bi-level positive airway pressure (CPAP/BIPAP) used solely for sleep-disordered breathing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Mortality at Day 28 | Randomization through Day 28
  All-cause mortality at Day 28

SECONDARY OUTCOMES:
Mortality at Days 60 and 90 | Randomization through Day 60 and Day 90
  All-cause mortality at Days 60 and 90
Number of ventilator-free days | Randomization through Day 28
  Number of ventilator-free days through Day 28
Improvement in oxygenation | Randomization to Day 2, Day 4, Day 6, Day 14, Day 28
  Improvement in oxygenation at Day 2, 4, 6, 14, and 28 compared to Baseline, as assessed by PaO2/FiO2
SOFA score at Day 28 | Randomization to Day 28
  SOFA score at Day 28 compared to Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics
Locations (1):
- Fresno Community Hospital, Fresno, California, United States